CLINICAL TRIAL: NCT03655366
Title: Investigation of Behaviour by Dogs Prior to Human Epileptic Seizures and Potential Underlying Mechanisms. Part 1:International Inventory of Seizure Dogs
Brief Title: Epidogs International Inventory of Seizure Alert Dogs
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: EC/2017/0934
Record Dates: First submitted 2017-11-07; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Epilepsy
Keywords: epilepsy; seizures; seizure alert dogs; seizure response dogs; assistance dogs
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dog owners with epilepsy: Epilepsy patients that own one or more dogs.
  Interventions: Other: Questionnaire for Dog owners
- Training organisations: Trainers of seizure response and seizure alerting dogs.
  Interventions: Other: Questionnaire for Dog trainers

INTERVENTIONS:
Other: Questionnaire for Dog owners — Questionnaire directed to epileptic patients, parents of epileptic children and legal representatives of epileptic patients with intellectual disabilities. It includes questions about demographics, epilepsy diagnosis, seizures, the behavior of their dogs around the time they have a seizure and a validates scale to measure dog personality traits.
  Groups: Dog owners with epilepsy
Other: Questionnaire for Dog trainers — Questionnaire for seizure response and seizure alert dog trainers including information on number of active working dogs, dog demographic information and selection criteria, the type of patient inclusion criteria they use, training methods used.
  Groups: Training organisations

SUMMARY:
This international research project looks at the reliability of canine seizure alerting behaviour in epilepsy patients. In the first stage an international database to identify the size and composition of the population of seizure alerting dogs has been created.

DETAILED DESCRIPTION:
The size and composition of the population of seizure alerting dogs is still widely unknown, particularly the population of non-trained alerting dogs. Previously published studies have focused on anecdotal reports, single case studies, or small samples of the population. Some studies do not make a clear distinction between response and alert dogs and/or include only one type of alerting dogs. The objective of this study is to create an international alerting dog database including trained Seizure Alert Dogs (SADs), spontaneously alerting Seizure Response Dogs (SRDs) and spontaneously alerting pet dogs. This information will be used to select a representative sample of the population for subsequent work packages and to perform a descriptive analysis of the population of alerting dogs in and international context. For the database, two questionnaires will be developed: one will be directed to SDR and SAD trainers and a second one to epilepsy patients owning a dog.

Questionnaires

The Trainer Questionnaire will be sent to training organisations via email and will request the following information:

* Number of active working dogs.
* Dog demographic information and selection criteria.
* The type of patient inclusion criteria they use
* Training methods used.
* For SRD that spontaneously started anticipating seizures: information about further training that may have been provided.

The questionnaire directed to epilepsy patients owning dogs will be accessible from our website and will collect the following information:

* Demographic information
* Information about the seizures
* Type of dog: SAD or spontaneously alerting SRD or pet dog
* Approximate date when the dog started alerting, if it's an untrained dog.
* Demographic information about the dog.
* Type of alerting behaviour.
* Monash Canine Personality Questionnaire refined (MCPQ-R): Defines 5 traits of dog personalities.
* The Monash Dog-Owner Relationship Scale (MDORS) ) that studies the perceived bond between the patient and the dog. It consists of 28 items with a score ranging from 1 to 5 that characterizes the emotional closeness, the dog-owner interaction and the perceive costs of dog ownership (Only for patients older than 18 year old)

Recruitment

Collaboration with epilepsy research groups has been stablished inside and outside the EU (Belgium, UK, US, Italy< Germany and Spain).

A systematic online search was performed to identify all SRD and SAD training organisations across the world. These organisations were contacted via email and telephone (see email example document) and asked to participate in the study by completing the trainer questionnaire and by distributing information about the study and an invitation to participate between their clients.

To reach epileptic owners of non-trained dogs that presumably alert, the following organisations were contacted:

* Epilepsy support organizations.
* Medical non-profit organisations
* Social media groups and forums.
* neurology departments and epilepsy centers

Milestones

* To create an international database of alerting dogs (SAD and spontaneously alerting SRD and pet dogs) to be used in subsequent work packages.
* Descriptive analysis of the population of alerting dogs and their owners.
* A description of the human-dog relationship between epileptic patients and their dog (separated according to whether the dog is one that alerts or not). A description of "Personality traits" of alerting and non-alerting dogs.

ELIGIBILITY:
Inclusion Criteria:

* Adults ( >18 years) diagnosed with epilepsy who live with a dog
* Children (< 18 years) that have been diagnosed with epilepsy and live with a dog; represented by the parents
* Epilepsy patients with intellectual disabilities that live with a dog; represented by their legal representative

Exclusion Criteria:

* Participants or their representative must be able to answer questions using our online questionnaire. They must sign the inform consent to access the questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dog owners (adults and children) with epilepsy
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Descriptive analysis of the population of owners of alerting and non-alerting dogs | Until October 2020
  Comparison of the responses from owners of alerting dogs and the responses of owners of non-alerting dogs in terms of type and frequency of seizures, presence or not od pre-ictal symptoms, etc.

SECONDARY OUTCOMES:
Differences in personality traits between alerting and non alerting dogs | Until October 2020
  Differences between the scores obtained in the MCPQ-R scale by alerting and non alerting dogs
Differences in human-dog bond between alerting and non alerting dogs | Until October 2020
  Differences between the scores obtained in the MDORS scale by alerting and non alerting dogs

CONTACTS AND LOCATIONS:
Overall Officials: Christel Moons, PhD, Study Director — Faculty of Veterinary Medicine, Ghent University
Locations (1):
- Department of Neurology - Ghent University Hospital, Ghent, Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dwyer, F., Bennett, P.C., Coleman, G.J., 2006. Development of the Monash Dog Owner Relationship Scale (MDORS). Anthrozoos 19, 243-256.
- [Background] Kirton A, Wirrell E, Zhang J, Hamiwka L. Seizure-alerting and -response behaviors in dogs living with epileptic children. Neurology. 2004 Jun 22;62(12):2303-5. doi: 10.1212/wnl.62.12.2303. PMID 15210902
- [Background] Ley, J.M., Bennett, P.C., Coleman, G.J., 2009a. A refinement and validation of the Monash Canine Personality Questionnaire (MCPQ). Appl. Anim. Behav. Sci. 116, 220-227
- [Background] Inter-rater and test-retest reliability of the Monash Canine Personality Questionnaire-Revised (MCPQ-R)
- See also: Website to access the questionnaires and the informed consents. — http://www.epidogsproject.net

DOCUMENTS (2):
  • Study Protocol (2017-06-24): https://cdn.clinicaltrials.gov/large-docs/66/NCT03655366/Prot_000.pdf
  • Informed Consent Form (2017-05-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT03655366/ICF_001.pdf